CLINICAL TRIAL: NCT00599885
Title: Comparison of Effects of Telmisartan and Valsartan on Neointima Volume in Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Associate professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TELLME; TELLME trial
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension; Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Coronary Artery Disease | interventions — Telmisartan; Valsartan

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: telmisartan
- 2 (Active Comparator)
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: telmisartan — telmisartan 40-80mg once per day for 8 months
  Arms: 1
Drug: valsartan — valsartan 80-160mg once per day for 8 months
  Arms: 2

SUMMARY:
People with diabetes mellitus are more prone to coronary heart disease, stroke, and peripheral vascular disease, and diabetes mellitus has been regarded as an independent risk factor for the progression of coronary artery disease. Several studies have been reported that diabetes increased the risk of cardiovascular mortality in both men and women. With the introduction of drug-eluting stents (DESs), the angiographic rates of restenosis at later months have reduced dramatically in several studies. However, even with DESs, diabetic patients showed increased rates of restenosis and late loss index compared with nondiabetic patients. Diabetes has been considered to be a predictor of poor prognosis after percutaneous coronary intervention with drug-eluting stents. Long-term clinical and angiographic outcomes after percutaneous coronary intervention (PCI) with drug-metal stents (DESs) have been demonstrated to be worse in diabetic patients compared with nondiabetic patients. In the era of DESs, no study has compared the effects of telmisartan and valsartan on neointima volume with intravascular ultrasound (IVUS) at 8 months after zotarolimus-eluting stent implantation in hypertensive type 2 diabetic patients. Telmisartan, which is well-known for its selective peroxisome proliferator-activated receptor (PPAR)-γ activity with its anti-inflammatory and antiproliferative properties, could be an appropriate therapeutic option for treating hypertensive diabetic patients with significant coronary artery diseases requiring stent implantation. In contrast, valsartan is an angiotensin receptor blocker with negligible PPAR-γ activity. Increasing interest remains in the identification of systemic pharmacological therapies to prevent coronary restenosis especially in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Gender eligible for study: both
* Hypertensive diabetic patients either previously diagnosed or newly found.
* Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 80 mmHg for newly found hypertensive patients.
* Fasting blood glucose ≥ 126 mg/dl or PP2 blood glucose ≥ 200 mg/dl for newly found diabetes.
* Patients with significant de novo coronary artery disease (diameter stenosis > 70%) requiring stent implantation (angina pectoris and/or exercise-induced ischemia).
* Patients with informed consent.

Exclusion Criteria:

* Acute ST-segment elevation myocardial infarction (MI), CTO lesions, left main lesions
* Diabetic patients with the use of thiazolidinediones within 3 months
* Previous history of PCI or bypass surgery
* Patients with any contraindications to the treatment of telmisartan or valsartan
* Pregnant or lactating patients
* Chronic alcohol or drug abuse
* Hepatic dysfunction
* Renal dysfunction
* Heart failure (EF < 50%)
* Expected life expectancy of < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Comparison of telmisartan and valsartan on neointima volume with IVUS at 8 months after zotarolimus-eluting stent implantation. | 8 month follow-up

SECONDARY OUTCOMES:
Comparison of telmisartan and valsartan on the levels of RBP-4 and inflammatory markers (hsCRP, IL-6, TNF-α, adiponectin). | 8 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Do-Sun Lim, MD, PhD, Study Chair — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Hong SJ, Choi SC, Ahn CM, Park JH, Kim JS, Lim DS. Telmisartan reduces neointima volume and pulse wave velocity 8 months after zotarolimus-eluting stent implantation in hypertensive type 2 diabetic patients. Heart. 2011 Sep;97(17):1425-32. doi: 10.1136/hrt.2011.225193. Epub 2011 Jun 23. PMID 21700754